CLINICAL TRIAL: NCT06815731
Title: Multicenter Study on the Correction of Prolapse Via Laparoscopy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-3-8-HCUVA
Record Dates: First submitted 2025-01-30; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Pelvic Floor Disorders
MeSH Terms: conditions — Pelvic Floor Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- lateral laparoscopic suspension (LLS) (Experimental)
  Interventions: Procedure: lateral laparoscopic suspension (LLS)
- Sacropexy without posterior mesh fixation on the puborrectalis muscle (Active Comparator)
  Interventions: Procedure: Sacropexy without posterior mesh fixation on the puborrectalis muscle

INTERVENTIONS:
Procedure: lateral laparoscopic suspension (LLS) — lateral laparoscopic suspension (LLS)
  Arms: lateral laparoscopic suspension (LLS)
Procedure: Sacropexy without posterior mesh fixation on the puborrectalis muscle — Sacropexy without posterior mesh fixation on the puborrectalis muscle
  Arms: Sacropexy without posterior mesh fixation on the puborrectalis muscle

SUMMARY:
In the laparoscopic lateral suspension (LLS) technique, the fixation of the mesh as a prosthetic element for correcting anterior apical vaginal prolapse at the level of the dome or uterus can offer anatomical and functional results that are not inferior to those of the conventional surgical technique, minimize possible intraoperative complications and facilitate the specific learning curve of sacropexy.

DETAILED DESCRIPTION:
In the laparoscopic lateral suspension (LLS) technique, the fixation of the mesh as a prosthetic element for correcting anterior apical vaginal prolapse at the level of the dome or uterus can offer anatomical and functional results that are not inferior to those of the conventional surgical technique, minimize possible intraoperative complications and facilitate the specific learning curve of sacropexy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Stage II- IV primary or recurrent prolapse affecting the anterior or middle vaginal compartment with or without minimal posterior defect (Stage I) according to the POP-Q.

Exclusion Criteria:

* History of abdominal prolapse reconstructive surgery.
* History of prolapse reconstructive surgery with vaginal meshes.
* Stage I according to the POP-Q classification or asymptomatic prolapse.
* Medical contraindication for general anaesthesia.
* Patient preference for vaginal surgical treatment.
* Patient does not wish to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 181 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Distress Inventory | up to 12 months
  Pelvic Organ Prolapse Distress Inventory (POPDI-6) Scores range between 0 and 24 for the POPDI-6
Colorectal-Anal Distress Inventory | up to 12 months
  Colorectal-Anal Distress Inventory (CRADI-8) Scores between 0 and 32 for the CRADI-8
Urinary Distress Inventory | up to 12 months
  Urinary Distress Inventory (UDI-6) Scores between 0 and 24 for the UDI-6.
Number of patients with symptomatic failure | up to 12 months
  Number of patients with symptomatic failure , defined as a positive response (accompanied by any degree of discomfort) to the following question on the validated questionnaire regarding prolapse symptoms (PFDI-20): "Do you usually have a bulge or something falling out that you can see or feel in your vaginal area?"

SECONDARY OUTCOMES:
Intestinal and pain symptoms | up to 12 months
  Subjective or functional success is defined as an improvement of ≥15 points per domain (the minimally important difference) or a decrease in the total score of 45 points (the minimally important difference). The PISQ-2 questionnaire has a score range between 0 and 48, and a difference ≥ 6 points is considered a minimally important difference.
Anatomical result | up to 12 months
  Anatomical results are defined as any POP-Q measurement below the hymen.
  Anatomical variables of prolapse: POPQ classification :
  * Anterior compartment: Aa, Ba
  * Middle compartment: C or D
  * Posterior compartment: Ap, Bp

CONTACTS AND LOCATIONS:
Locations (1):
- HCUVA, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No